CLINICAL TRIAL: NCT06705829
Title: Comparative Evaluation of the Performance of Different Thromboplastin Reagents on Prothrombin Time and Factorial Assays in Situations of Isolated Extrinsic Pathway Factor Deficiency or Liver Damage.
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: IV-0196
Record Dates: First submitted 2024-11-19; First posted 2024-11-26 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Hemorrhagic Disorders; Extrinsic Pathway Factor Deficiency; Hepatocellular Insufficiency With Coagulopathy
Keywords: Thromboplastin sensitivity; Prothrombin time
MeSH Terms: conditions — Hemorrhagic Disorders | interventions — Prothrombin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma samples obtained after centrifugation of whole blood samples collected in citrated tubes at 2500 g for 10 minutes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hepatocellular insufficiency with coagulopathy: Patients with an hepatocellular insufficiency generally associated with coagulopathy (with an intensity proportional to the degree of hepatic impairment).
  Interventions: Biological: Prothrombin

INTERVENTIONS:
Biological: Prothrombin — Comparison of prothrombin time results obtained with the different thromboplastins reagent for subgroup (extrinsic pathway factor and for those with hepatocellular insufficiency) by a regression line and a Bland-Altman representation.
  Comparison of extrinsic pathway factor assays obtained with the different thromboplastins reagent for each subgroup by a regression line and a Bland-Altman representation.
  Evaluation and determination of the sensitivity of the prothrombin time according to the activity rate obtained for each factor (for each reagent).

SUMMARY:
Primary purpose :

Compare the sensitivity of several thromboplastin reagents of various origins to prothrombin time and factor II, V, VII and X assays in two different populations of patients :

* Patients with an isolated extrinsic pathway deficiency (acquired or congenital) of factor II or V or VII or X.
* Patients with an hepatocellular insufficiency generally associated with coagulopathy (with an intensity proportional to the degree of hepatic impairment).

Results of this work should improve knowledge of sensitivity of the screening test represented by the prothrombin time, depending on the origin of thromboplastin reagent used, in relation with coagulopathies mentioned above, as well as the performance of factors II, V, VII, X assays. This work would help to choice of the most suitable reagent for the needs of each hemostasis laboratory/center.

ELIGIBILITY:
Inclusion criteria :

* Plasma samples from patients addressed to the laboratory of the Strasbourg University Hospital (Strasbourg France) collected and anonymized after completion of the routine testing.
* Patient with an isolated or combined extrinsic pathway factor deficiency (factor II, V, VII, X).

Exclusion criteria :

* Patient treated with an oral anticoagulant treatment.
* Patient treated with a parenteral anticoagulant treatment (apart from therapeutic dosages of unfractionated heparin and low molecular weight heparin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with an isolated (acquired or congenital) extrinsic pathway factor deficiency or with an hepatocellular insufficiency associated with a coagulopathy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-14 (Actual); Primary Completion 2024-12-14 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of the sensitivity of several thromboplastin reagents on prothrombin time and factor II, V, VII and X assays | 18 months
  Comparison of prothrombin time results obtained with the different thromboplastins reagent for subgroup (extrinsic pathway factor and for those with hepatocellular insufficiency) by a regression line and a Bland-Altman representation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg - Laboratoire de Virologie, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided